CLINICAL TRIAL: NCT04737057
Title: Clinical Efficiency and Child's Behavior of Hall Versus SDF Techniques in the Management of Carious Primary Molar:
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Lamiaa Saeed Ahmed Elshiekh, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CairoU1234
Record Dates: First submitted 2021-01-20; First posted 2021-02-03 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Early Childhood Caries
Keywords: hall technique; Silver diamide fluoride; non invasive technique
MeSH Terms: interventions — silver diamine fluoride

STUDY DESIGN:
Masking Description: not possible, since interventions are different
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hall Technique (Active Comparator): The Hall Technique is a non-invasive treatment for decayed molar teeth. Decay is sealed under preformed (stainless steel) crowns, avoiding injections and drilling. It is one of a number of biologically orientated strategies for managing dental decay
  Interventions: Procedure: SDF; Procedure: Hall technique
- SDF (Experimental): a clear liquid that combines the antibacterial effects of silver and the remineralizing effects of fluoride, is a promising therapeutic agent for managing caries lesions in young children and those with special care needs
  Interventions: Procedure: SDF; Procedure: Hall technique

INTERVENTIONS:
Procedure: SDF — Apply this topical medication through : 1)Dry with a gentle flow of compressed air to decayed tooth surfaces. 2) Bend micro sponge brush to remove excess liquid before application apply SDF directly to only the affected tooth surface. 3) Apply the SDF material 4)Dry with a gentle flow of compressed air for at least one minute. and Remove excess SDF with gauze
  Other Names: Silver Diamine Fluoride
Procedure: Hall technique — this technique is performed through :1) Orthodontic separator being stretched between two pieces of floss, then placed between the contact points of primary molars (for five days.) 2)The correct size of crown will not impinge on the teeth on either side, and a slight 'spring back' will be felt when the PMC is gently pushed up to (but not through) the contact points and the PMC has been filled with a Riva self-cure capsule cement, extruded cement is quickly wiped away and the child is asked to keep biting on the crown for two minutes, until the cement is set, to prevent 'spring back' of the PMC from the fully seated position

SUMMARY:
This study will compare two non- invasive treatment options: Hall technique and 38% Silver diamine fluoride. Both are methods used to create a more favorable environment without removal of caries leading to the arrest of the progression of demineralization process and restoring the function of the diseased molars.

DETAILED DESCRIPTION:
Dental caries, also known as tooth decay, it can occur in primary teeth in early childhood, is formed through interaction between acid-producing bacteria and carbohydrate. The caries develops in both the crowns and roots of teeth. Progress of caries depended on the lifestyle of the child (as high numbers of cariogenic bacteria, inadequate salivary flow, insufficient fluoride exposure and poor oral hygiene). To avoid this disease should follow the proper oral hygiene and improve lifestyle . A lot of methods found to treatment the decayed tooth - like; Hall technique and Silver diamine fluoride The first report on the Hall Technique published in 2007 by a general dental practitioner from Aberdeen/Scotland, Dr. Norna Hall. Dr. Hall used PMCs to restore carious primary molars rather than using the standard technique, placed them using a simplified method2

Previous studies have recommended that Silver diamine fluoride (SDF) solution would exert a preventive result in managing early childhood caries ECC. However, no well-designed clinical trials have yet been performed to study the effect of SDF on caries prevention. the objective is useful in arresting early childhood caries (ECC)

ELIGIBILITY:
Inclusion Criteria:

1. Age: From 4 to 6 years
2. Caries in primary molars within enamel / dentin without pulp disease

Exclusion Criteria:

1. Presence of signs and symptoms of necrosis
2. Root caries
3. Spontaneous pain

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Child's behavior | immediately after the procedure
  evaluate the Child's behavior by Frankl scale (FS) through Scores (1-2-3-4) ,(higher scores mean a better outcome)

SECONDARY OUTCOMES:
Canine overbite | one year
  measure the canine over bite discrepancy by Boley Gauge by Millimeter
Arresting caries in SDF | one year
  assess caries activity according to International Caries Detection and Assessment System (ICDAS) through Codes 0-1-2-3-4-5-6 ,( higher scores mean a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: gihan abo el neil, professor, Study Chair — Cairo University; ahmed alkhadem, assistant professor, Study Director — Cairo univeristy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: 2 years